CLINICAL TRIAL: NCT02400229
Title: Diagnostic Imaging Strategies for Patients With Stable Chest Pain and Intermediate Risk of Coronary Artery Disease: Comparative Effectiveness Research of Existing Technologies) - A Pragmatic Randomised Controlled Trial of CT Versus ICA
Brief Title: Diagnostic Imaging Strategies for Patients With Stable Chest Pain and Intermediate Risk of Coronary Artery Disease
Acronym: DISCHARGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marc Dewey, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: EA1/294/13; EC-GA 603266 (Other Grant/Funding Number: European Commission); Z 5 - 22462/2 - 2014-001 (Other: German Federal Office for Radiation Protection)
Record Dates: First submitted 2015-01-15; First posted 2015-03-27 (Estimated); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; stable chest pain; intermediate pretest probability; pragmatic randomised controlled trial; coronary computed tomography; angiography; invasive coronary angiography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computed Tomography Angiography (CTA) (Experimental): Computed Tomography Angiography including coronary calcium scoring and coronary computed tomography angiography
  Interventions: Procedure: Computed tomography angiography (cardiac CT)
- Invasive coronary angiography (ICA) (Active Comparator): Invasive coronary angiography
  Interventions: Procedure: Invasive coronary angiography (ICA)

INTERVENTIONS:
Procedure: Computed tomography angiography (cardiac CT) — Clinical management/treatment decisions based on cardiac computed tomography including coronary calcium scoring and coronary computed tomography angiography
  Arms: Computed Tomography Angiography (CTA)
Procedure: Invasive coronary angiography (ICA) — Clinical management/treatment decisions based on invasive coronary angiography
  Arms: Invasive coronary angiography (ICA)

SUMMARY:
The primary hypothesis is that computed tomography (CT) is superior to invasive coronary angiography (ICA) concerning the primary endpoint MACE (MACE = major adverse cardiovascular event; defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke) after a maximum follow-up of 4 years, in other words, that CT will result in a significantly lower rate of MACE. Secondary outcomes include MICE (MICE = minor cardiovascular events), procedural complications, cost-effectiveness, radiation exposure, cross-over to CT or ICA, gender differences, and health-related quality of life.

DETAILED DESCRIPTION:
The primary objective of this prospective pragmatic randomised controlled trial (PRCT) in 3546 patients is to evaluate the possible superiority of a CT-based patient management over an ICA-based management strategy in stable chest pain patients with intermediate pretest probability (10-60%) of coronary artery disease. The primary outcome measure is the occurrence of MACE (MACE = major adverse cardiovascular events; defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke) after a maximum follow-up of 4 years after CT or ICA. Secondary outcomes include health related quality of life, cost-effectiveness, cross-over to ICA/CT. Procedural complications are classified into major and minor. Major procedural complications are a composite end-point and include death, nonfatal stroke, nonfatal myocardial infarction, and further complications prolonging hospitalization by at least 24 hrs,as well as dissection (coronary, aorta), cardiogenic shock, cardiac tamponade, retroperitoneal bleeding, cardiac arrhythmia (ventricular tachycardia, ventricular fibrillation), cardiac arrest. Possible minor procedural complications: Hematoma at the puncture site, secondary bleeding at the puncture site, bradycardia, angina without infarction, allergoid contrast agent reaction, stent migration, hypotension requiring treatment, headache, hyperthyreodism, skin tissue and nerve injuries, extravasate, cardiac arrhythmia, contrast-induced nephropathy (CIN), infections, femoral arterial occlusion (or arterial access vessel) or dissection, new requirement for dialysis, DVT/pulmonary embolism, closure or injury of vessels, injury of the heart (e.g. valve or myocardium), , perforation, gastrointestinal bleeding, genital-urinary bleeding, other major bleeding, red blood cell (RBC)/whole blood transfusion, twisting or rupture of the catheter part, other equipment mishaps (e.g. retained foreign body guidewire fracture), development of arterio-venous fistula(s), development of pseudo aneurysm at puncture site, dissection (except coronary dissection), permanent edema (e.g. due to lymphatic congestion at puncture site), embolisation of central or peripheral vessels due to thromboembolis, acute closure of coronary vessels, stent infection, heart failure, wrong patient or wrong procedure and other.

This study is a European multicentre study conducted at 26 clinical centres in 16 European countries and is methodologically based on the single-centre CAD-Man trial conducted by Charité (NCT00844220). The pragmatic approach of the study ensures generating practical and usable outcomes for clinical decision-making according to comparative effectiveness research methodology.

In a preceding pilot study, data for cost-effectiveness analyses and image-quality analyses are collected and methods are defined for implementation in the main PRCT. Also appropriate instruments for health related quality of life are being chosen.

DISCHARGE receives funding from the 7th Framework Programme of the European Commission (EC-GA 603266).

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected coronary artery disease with stable chest pain and intermediate pretest probability (10-60%) of CAD referred for conventional coronary angiography.

"Stable chest pain" defined as not:

* being acute (= first appearance within the last 48 hours) or
* instable (= a) first appearance with at least Canadian Cardiovascular Society Angina Grading Scale (CCS) Class III, b) progredient with at least 1 CCS Class to at least CCS Class III or, now at rest for at least 20 min) angina pectoris
* Patients at least 30 years of age
* Written informed consent

Exclusion Criteria:

* Patients on hemodialysis
* No sinus rhythm
* Pregnancy
* Any medical condition that leads to the concern that participation is not in the best interest of health (e.g., extensive comorbidities)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3546 (Estimated)
Dates: Start 2015-10-03 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Event | 1 minute after randomisation to CT/ICA diagnostic procedure and during follow-up
  Composite endpoint: major adverse cardiovascular event (MACE); defined as at least one of the following: cardiovascular death, nonfatal myocardial infarction, and nonfatal stroke.

SECONDARY OUTCOMES:
Likelihood of receiving coronary intervention in different European countries | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  Likelihood of receiving coronary intervention and extent of Coronary Artery Disease (CAD) in dependence of socioeconomic status and the likelihood of receiving further intervention within two months after the initial intervention in different European countries.
Rates of percutaneous coronary intervention and use of intracoronary techniques different European countries | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  Composite outcome: Rates of Percutaneous Coronary Intervention (PCI) and use of intracoronary techniques such as Fractional Flow Reserve (FFR), Optical Coherence Tomography (OCT), Intravascular Ultrasound (IVUS) within two months after the initial intervention in different European countries.
Patient management in different European countries | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  Recommended and actually performed management based on Computed Tomographic Angiography (CTA) and Invasive Coronary Angiography (ICA) results in different countries adjusted for the extent of ischemia within two month after the initial test randomised to.
Follow-up strategies in different European countries | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  Composite outcome: Adherence to follow-up in different countries and according to prevalence of CAD as well as risk factors and socioeconomic status and most likely way of conduct of follow-up data gathering in different countries (phone interviews, letter reply, email).
European differences in occurrence and extent of Coronary Artery Disease in regards to city versus rural lifestyle | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  European differences in occurrence and extent of Coronary Artery Disease in regards to city versus rural lifestyle
European and local differences in patient consent of sites | at baseline, 1-year follow-up and final follow-up up to a max of 4 years
  European and local differences in patient consent of sites
Comparison in the Coronary Computed Tomographic Angiography and Invasive Coronary Angiography group:Occurrence of Minor Adverse Cardiovascular Events | 1 minute after randomisation to CT/ICA diagnostic procedure and during follow-up
  Occurrence of minor adverse cardiovascular events (MICE): coronary revascularisation, peripheral artery revascularisation, hospitalisation for angina pectoris, emergency department visit for angina pectoris, transient ischemic attack, congestive heart failure.
Comparison in the Computed Tomography Angiography and Invasive coronary Angiography group: Percutaneous Coronary Intervention and Coronary Artery Bypass Graft | during the CTA/ICA examination, up to 48h after hours after the final procedure related to the test randomized to, 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Rates of Percutaneous Coronary Intervention and Coronary Artery Bypass Graft (CABG) performed within 2 months following Computed Tomography Angiography and Invasive Coronary Angiography (defined as: related to these tests) and more than 2 months after CTA and ICA until follow-up (unrelated to these tests).
Comparison in the Computer Tomography Angiography and Invasive Coronary Angiography group: Rates of patients on dialysis | during the CTA /ICA examination, up to 48h after hours after the final procedure related to the test randomized to, 1-year follow-up and final follow-up to a max of 4 years
  Comparison in the CTA and ICA group: Rates of patients on dialysis
Comparison in the Computer Tomography Angiography and Invasive Coronary Angiography group: Rate of coronary anatomical anomalies | during the CTA /ICA examination, up to 48h after hours after the final procedure related to the test randomized to, 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Rate of coronary artery anomalies (benign and malignant) and rate of myocardial bridging seen on CTA and ICA and the clinical implications of these at follow-up as well as influence on Major Adverse Cardiovascular Events (MACE) and MICE
Comparison in the computer tomography angiography and invasive coronary angiography group: Rates of patients undergoing further cardiac diagnostics | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Composite outcome: Rates of patients undergoing further cardiac diagnostics, such as additional CT or ICA, Electrocardiography (ECG), Exercise ECG, Echo, Stress Echo, Magnetic Resonance Imaging (MRI) within 2 months following CT and invasive coronary angiography (defined as: related to these tests) and more than 2 months after CT and invasive coronary angiography until follow-up (unrelated to these tests).
Comparison in the computer tomography angiography and invasive coronary angiography group: Rates of coronary interventions | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Rates of coronary interventions within 2 months following CT and ICA (defined as: related to these tests) and more than 2 months after CT and ICA until follow-up and recurrent angina leading to hospitalisation.
Analysis of the influence of prior computer tomography angiography on invasive coronary angiography and percutaneous coronary intervention | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Analysis of influence of prior CT on ICA and PCI in terms of duration, radiation exposure, amount of contrast agent used for ICA.
Comparison of cumulative contrast agent amount in the two arms | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Comparison of cumulative contrast agent amount in the two arms
Comparison in the computer tomography angiography and invasive coronary angiography group: Number/proportion of patients undergoing coronary revascularization | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Composite outcome: Compared with ICA, CTA will be associated with a lower rate of coronary revascularisation, but on a per-procedure basis, revascularisation will be more complete. Performance of revascularisation will differ between the randomised groups.
Comparison in the computer tomography angiography and invasive coronary angiography group: Distribution in the mode of revascularization: percutaneous coronary intervention vs. coronary artery bypass graft | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow up to a max of 4 years
  Comparison in the CTA and ICA group: Distribution in the mode of revascularisation: PCI vs. CABG.
Comparison of Quality of Life between treatment regimens. | at 1-year follow-up and final follow-up to a max of 4 years
  Comparison of Quality of Life between the following treatment regimens using adherence to therapy recommendation as covariate: optimal medical therapy in general in combination with risk factor modification vs. oral statin intake in combination with risk factor modification.
Geographical distribution of risk factors for Major Cardiovascular Events and Minor Cardiovascular Events and other events | at 1-year follow-up and final follow-up to a max of 4 years
  Geographical distribution of risk factors for MACE and MICE, cardiovascular events and cardiac events (cardiac and non-cardiac death, stroke, myocardial infarction, unstable angina pectoris, re-revascularisation and first revascularisation) in the European Union (EU) and comparison of European countries.
Extent of Coronary Artery Disease | at 1-year follow-up and final follow-up to a max of 4 years
  Extent of CAD in dependence of patients' socioeconomic status (income, education, occupation, job situation, gender)
Time from randomisation to Invasive Coronary Angiography in both groups | at 1-year follow-up and final follow-up to a max of 4 years
  Time from randomisation to Invasive Coronary Angiography in both groups.
Time from randomisation to first coronary revascularisation in both groups | at 1-year follow-up and final follow-up to a max of 4 years
  Time from randomisation to first coronary revascularisation in both groups
Completeness of revascularisation for Percutaneous Coronary Intervention single vessel vs multivessel Percutaneous Coronary Intervention and Coronary Artery Bypass Graft; stent use (bare metal vs drug eluting) | at 1-year follow-up and final follow-up to a max of 4 years
  Completeness of revascularisation (i.e. no. of vessels treated vs. number of vessels affected by > 50% stenosis); for Percutaneous Coronary Intervention single vessel vs multivessel Percutaneous Coronary Intervention and Coronary Artery Bypass Graft; stent use (bare metal vs drug eluting).
Information on surgical procedures i.e. isolated Coronary Artery Bypass Graft, Coronary Artery Bypass graft with valve replacement, Coronary Artery Bypass Graft with aortic surgery | at 1-year follow-up and final follow-up to a max of 4 years
  Information on surgical procedures i.e. isolated Coronary Artery Bypass Graft, Coronary Artery Bypass graft with valve replacement, Coronary Artery Bypass Graft with aortic surgery.
Comparison in the Computer Tomography Angiography and Invasive Coronary Angiography group: procedures and outcomes in relation to age | at 1-year follow-up and final follow-up to a max of 4 years
  Comparison in the Computer Tomography angiography and Invasive Coronary Angiography group: procedures and outcomes in relation to age.
Comparison in the Computer Tomography Angiography and Invasive Coronary Angiography group: procedures and outcomes in relation to body mass index and obesity | at 1-year follow-up and final follow-up to a max of 4 years
  Comparison in the Computer Tomography Angiography and Invasive Coronary Angiography group: procedures and outcomes in relation to body mass index and obesity.
Reduction of angina pectoris intensity | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Reduction of angina pectoris intensity (measured on a 0-10 scale, at baseline, first and final follow up, max 4 years) in the two arms and in the subgroup of a) patients with significant stenosis (on CTA or ICA) and with or without relevant myocardial ischemia that was or was not revascularised by PCI or CABG; b) patients without significant stenosis (on CT or ICA) and with or without non-coronary or non-cardiac finding potentially explaining the chest discomfort; in patients who underwent PCI versus patients who received optimal medical therapy and risk factor modification alone (matched analysis for the extent of CAD and imaging ischemia).
Validation of different questionnaires to predict Major and Minor Adverse Cardiac Events | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Validation of the Rose Angina questionnaire including pain scale and the InterHeart Risk Score (IHRS) to predict MACE and MICE in both arms.
Occurrence of adverse events due to medication | during the procedure or within 48 hours post last related procedure
  Composite outcome: Adverse events due to nitroglycerin, beta-blockers, contrast agent and other medication applied during CTA and ICA (allergic reactions, hypotension, headache, hyperthyroidism).
Occurrence of adverse events related to venous or arterial puncture | during the procedure or within 48 hours post last related procedure
  Composite outcome: Adverse events related to venous or arterial puncture: skin tissue and nerve injuries, bleedings: due to puncture of vessel, due to use of anticoagulants, at site of puncture (hematoma), extravasate.
Occurrence of cardiac arrhythmia | during the procedure or within 48 hours post last related procedure
  Occurrence of cardiac arrhythmia
Rates of contrast-induced nephropathy | up to 48h after hours after the final procedure related to the test randomised to
  Rates of contrast-induced nephropathy (CIN) adjusted for the frequency of creatinine follow-up testing performed in the two groups.
Infections | during the procedure or within 48 hours post last related procedure
  Infections
Influence of experience of examiners on events | during the procedure or within 48 hours post last related procedure
  Correlation of the experience (in years) of the CT and ICA examiner with procedural events, duration of the exams (in min), contrast agent amount (in ml) used for diagnosis and intervention (if done), and exposure of radiation (in mSv).
Comparison of occurrence of procedural complications related to Invasive Coronary Angiography | during the procedure or within 48 hours post last related procedure
  Composite outcome: Comparison of a) outpatient vs inpatient ICA for procedural complication rates after adjusting for risk factors for such events,b) femoral vs radial approach ICA, and c) different closure devices vs. manual compression and of frequency of interventions, results, patients acceptance and d) procedural differences, for instance bed rest time after intervention, and influence on procedural events.
Procedural complications related to Invasive Coronary Angiography | during the procedure or within 48 hours post last related procedure
  Composite outcome: Complications related to ICA: Femoral arterial occlusion (or arterial access vessel) or dissection, Cardiac arrhythmia, closure or injury of vessels, injury of the heart (e.g. valve or myocardium) , twisting or rupture of the catheter or parts of the catheter consecutive surgical removal, development of arteria-venous fistulas, development of a pseudo aneurysm at puncture site, permanent edemas, embolisation of central or peripheral vessels due to thromboembolism.
Procedural complications during or after revascularisation | during the procedure or within 48 hours post last related procedure
  Complications during or after revascularisation, for instance acute closure of coronary vessels, angina pectoris, stent migration, loss of stent and consecutive closure of vessels, stent infection.
Occurrence of other adverse events and serious adverse events in the Invasive Coronary Angiography group | during the procedure or within 48 hours post last related procedure
  Composite outcome: Occurrence of other adverse events (AEs) and serious adverse events (SAEs) such as heart failure, cardiogenic shock, cerebrovascular accident (CVA)/Stroke, hemorrhagic stroke, new requirement for dialysis, deep vein thrombosis/pulmonary embolism, cardiac tamponade, perforation, retroperitoneal bleeding, gastrointestinal bleeding, genital-urinary bleeding, major bleeding, red blood cell (RBC)/Whole blood transfusion, other equipment mishaps (e.g. retained foreign body guidewire fracture), wrong patient or wrong procedure
Comparison of incidental findings in Computed Tomography Angiography and Invasive Coronary Angiography group and potential benefits and harms of findings Analysis of prevalence non-coronary cardiac and non-cardiac causes of symptoms | during CTA and ICA examination, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a max of 4 years
  Analysis of prevalence of a) non-coronary cardiac causes of symptoms (such as aortic dissection, valve disease, pericarditis) or b) non-cardiac causes of symptoms (such as thrombus, pulmonary embolism, pleural effusion, pneumonia, hiatal hernia).
Comparison of incidental findings in both arms and potential benefits and harms of findings:Influence of non-coronary cardiac and non-cardiac findings on Major Adverse Cardiac Events, non-cardiac events and Quality of Life | during CTA and ICA examination, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a max of 4 years
  Influence of non-coronary cardiac and non-cardiac findings on MACE, non-cardiac events and Quality of Life (QoL).
Comparison of incidental findings in Computed Tomography Angiography and Invasive Coronary Angiography group and potential benefits and harms of findings: Rate for malignancy in nodules seen on Computed Tomography Angiography | during CTA and ICA examination, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a max of 4 years
  Rate for malignancy in nodules seen on CT (reference standard: biopsy results, Positron Emission Tomography (PET) findings, or progression versus no change or regression on follow-up CT.
Comparison of incidental findings in Computed Tomography Angiography and Invasive Coronary Angiography group and potential benefits and harms of findings | during CTA and ICA examination, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a max of 4 years
  Accuracy of the parsimonious lung cancer risk prediction tool by McWilliams et al. for probability assessment of malignancy in lung nodules found in comparison to the above combined reference standard
Comparison of incidental findings in Computed Tomography Angiography and Invasive Coronary Angiography group and potential benefits and harms of findings: Rate of death from cancer in both groups | at 1-year follow-up and final follow-up to a maximum of 4 years
  Rate of death from cancer in both groups
Comparison of incidental findings in Computed Tomography Angiography and Invasive Coronary Angiography group and potential benefits and harms of findings:Rates of unnecessary follow-up procedures | at 1-year follow-up and final follow-up to a maximum of 4 years
  Composite outcome: Rates of unnecessary follow-up procedures such as examinations, biopsies, or surgeries done based on non-coronary findings in the CTA and ICA group
Analysis of interobserver variability (site versus core lab) | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Analysis of interobserver variability (site vs. core lab) of reading for coronary stenosis and plaques on CTA and for coronary stenosis on ICA
Percent diameter stenosis correlation and agreement by both diagnostic tests in patients who underwent Invasive Coronary Angiography in the Computed Tomography Angiography group after positive or non-diagnostic findings | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Percent diameter stenosis correlation and agreement by Computed Tomography Angiography and Invasive Coronary Angiography in patients who underwent Invasive Coronary Angiography in the Computed Tomography Angiography group after positive or non-diagnostic findings.
Non-diagnostic Computed Tomography Angiography and Invasive Coronary Angiography | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Composite outcome: Non-diagnostic CTA and ICA: comparison of prevalence and patient as well as technical factors leading to such uninterpretable findings or exams that could not be conducted or completed.
Correlation between percent diameter stenosis | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Correlation between percent diameter stenosis by Computed Tomography with invasive Fractional Flow Reserve in patients who had Computed Tomography and Invasive Coronary Angiography done and correlation of non-invasively estimated Fractional Flow Reserve by Computed Tomography with invasive Fractional Flow Reserve after Computed Tomography/Invasive Coronary Angiography.
Prevalence of sinus node artery being a side branch of Left Coronary Artery or Right Coronary Artery | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Prevalence of sinus node artery being a side branch of Left Coronary Artery (LCX) or Right Coronary Artery RCA by core lab reading and the risk of CAD on CT and ICA as well as MICE and MACE.
Prevalence of left, intermediate, and right coronary distribution type | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Prevalence of left, intermediate, and right coronary distribution type by core lab and site reading and the risk of CAD (as significant) on CT and ICA at baseline and MICE and MACE.
Improvement of selection of distal coronary segments used for CABG-anastomosis by CT in comparison to ICA alone (especially heavy calcification detection) as assessed by the cardiac surgeons. | at 1-year follow-up and final follow-up to a maximum of 4 years
  Improvement of selection of distal coronary segments used for Coronary Artery Bypass Surgery-anastomosis by Computed Tomography in comparison to Invasive Coronary Angiography alone (especially heavy calcification detection) as assessed by the cardiac surgeons.
Relation of plaque characterisation and quantification by core lab and Major and Minor Adverse Cardiac Events at the two follow-up results | at 1-year follow-up and final follow-up to a maximum of 4 years
  Relation of plaque characterisation and quantification by core lab and MACE and MICE at the two follow-up results.
Image quality of Computed Tomography by core lab read and flow and concentration of contrast agent used intravenously | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Image quality of CT by core lab read and flow and concentration of contrast agent used intravenously
Coronary artery dimensions | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Coronary artery dimensions in patients in whom contraindications prevented the use of nitroglycerin for CTA versus patients who received nitroglycerin (measured as the diameter of the Left Marginal Artery (LMA), proximal Left Anterior descending artery (LAD), LCX and RCA), adjusted for gender and Body Surface Area (BSA).
Noise in Computed Tomography Angiography imaging | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Noise in CTA imaging and the factors it depends on for instance adherence vs non-adherence to scan protocol.
Factors that influence the image quality of Computed Tomography Angiography | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Factors that influence the image quality of CTA ( Body Mass Index (BMI), gender, origin of patient, 80, 100, 120, 135, 140 kV, different mA settings, number of detector rows, heart rate (maximum, minimum, and average during CT acquisition), and acquisition type.
Accuracy and agreement of RCADIA system | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
10-step Guide to cardiac CT | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Evaluation of the 10-step guide to cardiac CT
Semi-qualitative analysis | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Composite outcome: intensity, noise, signal to noise, contrast and signal to noise in some regions of interest (ROIs) (LV, RV segments 1,2,5,6,11 and levocardiography effect).
Qualitative analysis | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Composite outcome: levocardiography effect (scale 1 to 3) and LV, RV and segments 1,2,5,6,11 (scale 1 to 4).
Heart rate reduction achieved in Computed Tomography by the DISCHARGE betablocker protocol | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Heart rate reduction achieved in Computed Tomography by the DISCHARGE betablocker protocol
Heart rate reduction achieved in subgroups | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Composite outcome: Heart rate reduction achieved in subgroups of patients with contraindication to betablockers or no adherence to protocol where other doses or medications such as ivabradine or calcium channel blockers were used and in different patient groups (e.g., male versus female patients, >65 years and up to 65 years of age).
Heart rate reduction achieved with conscious sedation, if used, for Computed Tomography | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Heart rate reduction achieved with conscious sedation, if used, for CT.
Correlation of extent of Coronary Artery Disease and a high calcium score | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Composite outcome: Analysis of prevalence and extent of CAD in correlation to a high calcium score (CS), and exclusion of any CAD in correlation to a zero CS, potential of defining a threshold.
Characterisation of plaques | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  The characterisation of plaques (type and composition) by CT core lab in relation to cardiac risk factors.
Differences in plaque characteristics | during the Computed Tomography examination and up to 6 months after the Pragmatic Randomised Controlled Trial
  Composite outcome: Differences in plaque characteristics (type and composition) and analysis of potential influence by geographical origin of the patient, after adjustment for other cardiac risk factors.
Comparison of Computed Tomography Angiography and intracoronary techniques | during the Computed Tomography examination and up to 6 months after the pragmatic Randomised Controlled Trial
  Composite outcome: Correlation and agreement for plaque characterisation and quantification by CT in comparison to intracoronary techniques such as OCT and Intravascular ultrasound (IVUS) in patients who had both tests done.
Influence of statin treatment on plaque development | during the Computed Tomography examination and up to 6 months after the pragmatic Randomised Controlled Trial
  Risk factors for and influence of statin treatment on plaque progression or regression in patients who had follow-up cardiac CT done in the CT group.
Correlation of effective dose and the diagnostic portion of Invasive Coronary Angiography with weight and body-mass index of the patient. | during the Invasive Coronary Angiography examination, at 1-year follow-up and at final follow-up to a maximum of 4 years
  Correlation of effective dose and the diagnostic portion of Invasive Coronary Angiography with weight and body-mass index of the patient.
Correlation of effective dose of and contrast agent amount used for Invasive Coronary Angiography with severity of Coronary Artery Disease | during the Invasive Coronary Angiography examination, at 1-year follow-up and at final follow-up to a maximum of 4 years
  Correlation of effective dose of and contrast agent amount used for Invasive Coronary Angiography with severity of Coronary Artery Disease.
Rate of follow-up Invasive Coronary Angiographies and Percutaneous Coronary Interventions more than 2 months after initial Computed Tomography/Invasive Coronary Angiography and up to first and last follow-up | during the Invasive Coronary Angiography examination, at 1-year follow-up and at final follow-up to a maximum of 4 years
  Rate of follow-up Invasive Coronary Angiographies and Percutaneous Coronary Interventions more than 2 months after initial Computed Tomography/Invasive Coronary Angiography and up to first and last follow-up
Correlation of the number of projections for the right and left coronary artery with effective dose of Invasive Coronary Angiography | during the Invasive Coronary Angiography examination, at 1-year follow-up and at final follow-up to a maximum of 4 years
  Correlation of the number of projections for the right and left coronary artery with effective dose of Invasive Coronary Angiography
Rates of left ventriculography performed | during the Invasive Coronary Angiography examination, at 1-year follow-up and at final follow-up to a maximum of 4 years
  Rates of left ventriculography performed
Rates of planned cross-over from Computed Tomography to Invasive Coronary Angiography | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Rates of planned cross-over from CT to ICA after positive findings in CT within 2 month past initial procedure in accordance to management flow chart.
Comparison of cross-over patients (from Computed Tomography to Invasive Coronary Angiography) to non-cross-over-patients | up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Comparison of cross-over patients (from Computed Tomography to Invasive Coronary Angiography) to non-cross-over-patients.
Correlation of Computed Tomography Angiography and/or Invasive Coronary Angiography with the results of imaging ischemia tests | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Composite outcome: Correlation of CTA and/or ICA results with the results of imaging ischemia tests (stress echo, stress Single Photon Emission Computed Tomography (SPECT), stress Positron Emission Tomography (PET), MRI & stress MRI).
Correlation between imaging ischemia tests and invasive Fractional Flow Reserve if done | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Correlation between imaging ischemia tests and invasive Fractional Flow Reserve if done.
Rates of imaging ischemia tests recommended | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Rates of imaging ischemia tests recommended
Comparison of diagnostic accuracy of imaging ischemia tests | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Comparison of diagnostic accuracy of imaging ischemia tests (stress echocardiography, SPECT, stress MRI, and PET) for the detection of CTA- or ICA-defined CAD (up to 48h after final procedure related to the randomised test).
Comparison of imaging ischemia results with Computed Tomography Angiography and Invasive Coronary Angiography results for prediction of Major and Minor Cardiac Adverse Events | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Comparison of imaging ischemia results with Computed Tomography Angiography and Invasive Coronary Angiography results for prediction of Major and Minor Cardiac Adverse Events.
Correlation between imaging ischemia results and coronary stenosis as well as plaque composition and characterisation findings by Computed Tomography Angiography | at baseline, up to 48h after the final procedure related to the test randomised to, at 1-year follow-up and final follow-up to a maximum of 4 years
  Correlation between imaging ischemia results and coronary stenosis as well as plaque composition and characterisation findings by Computed Tomography Angiography.
Rate of revascularisations recommended and performed after Computed Tomography Angiography and positive or negative imaging ischemia tests in comparison to Invasive Coronary Angiography arm within two month after the initial test | at baseline, at 1-year follow-up and final follow-up to a maximum of 4 years
  13.2.1 Rate of PCI / CABG recommended and performed after CTA and positive or negative imaging ischemia tests in comparison to the ICA arm within two month after the initial test.
Correlation of the results of study- Computed Tomography Angiography, recommended imaging ischemia test and Invasive Coronary Angiography in patients with respective study course | at baseline, at 1-year follow-up and final follow-up to a maximum of 4 years
  Correlation of the results of study- CTA, recommended imaging ischemia test and ICA in patients with respective study course
Occurrence of procedural events in imaging ischemia testing | at baseline, at 1-year follow-up and final follow-up to a maximum of 4 years
  Occurrence of procedural events in imaging ischemia testing.
Correlation of intensity and reduction of angina pectoris | at baseline, at 1-year follow-up and final follow-up to a maximum of 4 years
  Correlation of intensity and reduction of Angina Pectoris (measured on a 0-10 scale, baseline, first and final follow up, max 4 years) with positive, unequivocal, and negative imaging ischemia test results in patients in both study arms; sub-study in patients with imaging ischemia follow-up examinations with an analysis of the correlation between changes in angina intensity and ischemia extent.
Analysis of patient acceptance ("preference questionnaire") of Computed Tomography Angiography and Invasive Coronary Angiography | at baseline, up to 48h after hours after the final procedure related to the test randomized to, 1-year follow-up and final follow-up to a max of 4 years
  Analysis of patient acceptance ("preference questionnaire") of CTA and ICA (and in those patients, who received both, which one was the preferred) as well as in the following subgroups: gender, patients without significant stenosis seen on the initial test randomised to, patients with significant stenosis seen on CTA and a) ICA not recommended or done e.g., because of imaging ischemia results or b) ICA done.
Patient acceptance of informed consent, preparation and procedural aspects of the test performed | at baseline, up to 48h after hours after the final procedure related to the test randomized to, 1-year follow-up and final follow-up to a max of 4 years
  Patient acceptance of informed consent, preparation, procedural aspects of the tests performed including an assessment of maximum pain during procedures measured using a pain scale and patient acceptance of the management recommendations in the two groups.
Effective radiation dose for Computed Tomography Angiography and Invasive Coronary Angiography | up to 48h after the final procedure related to the test randomised, at 1-year follow-up and final follow up to a max of 4 years
  Effective radiation dose (measures as dose length product and dose area product during CT [for coronary artery calcium score (CACS) and CTA] and ICA, respectively) used for CT and ICA and cumulative radiation dose in the two arms at different time points.
Reduction of radiation exposure by using coronary artery calcium score information | up to 48h after the final procedure related to the test randomised, at 1-year follow-up and final follow up to a max of 4 years
  Reduction of radiation exposure by using CACS information about the coronary artery position along the Z-axis to reduce the Z-axis coverage of the subsequent CTA according to the 10 Steps Guide to Success in Cardiac CT.
Comparison of radiation dose in Invasive Coronary Angiography and Computed Tomography Angiography: pilot study versus non-study patients | during Computed Tomography Angiography and Invasive Coronary Angiography Examination
  Comparison of radiation dose in ICA and CT: pilot study versus non-study patients
Validation of the coronary artery disease DISCHARGE and COME-CCT pre-test probability calculators | at 1-year follow-up and final follow-up to a maximum of 4 years
  Validation of the coronary artery disease DISCHARGE and COME-CCT pre-test probability calculators and comparison with other calculators (Diamond and Forrester, DiCAD, Duke clinical score) versus the reference standards (CTA or ICA) in the pilot study of DISCHARGE and the randomised trial.
Comparison of the ability of the DISCHARGE and COME-CCT pre-test probability calculators to predict Coronary Artery Disease indifferent genders | at 1-year follow-up and final follow-up to a maximum of 4 years
  Comparison of the ability of the DISCHARGE and COME-CCT pre-test probability calculators to predict CAD in men and women equally well in comparison to previous calculators.
Ability of the DISCHARGE and COME-CCT pre-test probability calculators to predict Coronary Artery Disease | at 1-year follow-up and final follow-up to a maximum of 4 years
  Ability of the DISCHARGE and COME-CCT pre-test probability calculators to predict CAD in patients without or with coronary artery calcium on CT using CTA or ICA as the reference standard in comparison to previous calculators.
Potential advantage of the DISCHARGE and COME-CCT calculators | at 1-year follow-up and final follow-up to a maximum of 4 years
  Potential advantage of the DISCHARGE and COME-CCT calculators in combination with the NIH chest discomfort guidelines to triage patients most effectively based on pretest probability in comparison to the DISCHARGE approach of CT including calcium scoring and CTA for management decision making about risk factor modification and revascularisation, respectively.
Predictive value of the DISCHARGE calculator in patients who could not be included in the trial due to their very low pre-test probability (<10%) | at 1-year follow-up and final follow-up to a max of 4 years
  Predictive value of the DISCHARGE calculator in patients with a very low pre-test probability (<10%) who could not be randomised but were sent with an indication for ICA that these patients, who are in a screening log of the study, actually have no CAD on ICA.
Predictive value of the DISCHARGE calculator | at 1-year follow-up and final follow-up to a max of 4 years
  Predictive value of the DISCHARGE calculator in patients with a high pre-test probability (>60%) who could not be randomised but were sent with an indication for ICA that these patients, who are in a screening log of the study, actually have a high risk of CAD on subsequent ICA.
Development and validation of a novel pre-test probability calculator | at 1-year follow-up and final follow-up to a maximum of 4 years
  Composite outcome: Development and validation of a novel pre-test probability calculator based on age, gender, symptoms, and cardiac risk factors and/or exercise ECG or imaging ischemia results of patients in DISCHARGE with CT and/or ICA results being the reference standard for the definition of CAD for this novel calculator; comparison of this novel calculator with the simple DISCHARGE pre-test probability calculator.
Ability of the DISCHARGE and COME-CCT calculators to predict Major and Minor Adverse Cardiac Events | at 1-year follow-up and final follow-up to a maximum of 4 years
  Ability of the DISCHARGE and COME-CCT (Collaborative Meta-analysis in Cardiac CT) calculators (used in the study and developed based on the study results) to predict MACE and MICE at both follow-up will be analysed.
Cost-Effectiveness Analysis | at 1-year follow-up and final follow-up to a max of 4 years
  In addition to the costs of CTA and ICA, we assess costs induced by complications caused by these diagnostic procedures. Those costs split up into costs for additional diagnostics and additional treatments necessary due to the occurrence of major cardiovascular adverse events. Therefore, number, type and severity of adverse events, caused by CTA and ICA will be evaluated as well as the type of treatment and if the treatment is conducted in an ambulant setting or requires hospitalisation.
Cost-Utility Analysis | at 1-year follow-up and final follow-up to a max of 4 years
  Comparison of the costs of an additional quality adjusted life year (QALY) gained by a correct diagnosis gained by using CTA or ICA.
Comparison of cost-effectiveness analysis and cost-utility analysis in different European countries | at 1-year follow-up and final follow-up to a max of 4 years
  All analyses including costs will be conducted separately for each country with a study center to enable us to conduct comparative analyses on an international level.
Average days off work per patient by clinical site during follow up | at 1-year follow-up and final follow-up to a max of 4 years
  Adverse events might lead to sick leave in patients, which is an important cost factor from the societal perspective. There will be an assessment of differences in sick leave in patients by clinical site.
Days in hospital per patient by clinical site during follow up | at 1-year follow-up and final follow-up to a max of 4 years
  Adverse events might lead to hospitalisation in patients. In addition to days off work, this is an important cost factor from the societal perspective. There will be an assessment of differences in hospitalisation in patients by clinical site.
Additional diagnostic tests during follow-up by clinical site | at 1-year follow-up and final follow-up to a max of 4 years
  Differences in adverse events might lead to a different use of diagnostic tests during the follow-up phase. Therefore, data about cost-effective differences in examinations, not being mandatory according to the study protocol, will be collected.
Additional treatments during follow-up by clinical site | at 1-year follow-up and final follow-up to a max of 4 years
  Differences in adverse events might lead to a different necessity of treatments during the follow-up phase. Therefore, data about cost-effective differences in treatments, not mandatory by study protocol, will be collected.
Pragmatic assessment of staff involvement time and material use - completion of questionnaires | up to a maximum of 2 years after completion of pilot study at all sites
  A pragmatic Case Report Form (CRF) for the assessment of staff involvement time and use of material was developed for the pilot study. The completion of questionnaires in different clinical sites will be assessed to evaluate this approach.
Differences in staff involvement time for Computed Tomography Angiography and Invasive Coronary Angiography in different clinical sites | up to a maximum of 2 years after completion of pilot study at all sites
  Differences in staff involvement time in different clinical sites will be assessed. Staff involvement time is one of the major cost drivers in health care systems.
Differences in consumption of materials in different clinical sites | up to a maximum of 2 years after completion of pilot study at all sites
  Different consumption of materials in different clinical sites will be assessed. Therefore we will use standardised prices for inter-site comparisons.
Comparison of population of pilot study between the different European clinical sites | up to a maximum of 2 years after completion of pilot study at all sites
  The pilot study is not a prospective randomised trial. Inclusion of patients with a pretest-likelihood greater than 60% was allowed due to retrospective calculation of pretest likelihood. Thus, the population in the pilot study differs from the population being included in the DISCHARGE main trial.
  As cost-effectiveness data will be calculated using data from the pilot study, controlling for age, gender, pretest-likelihood, and quality of live related parameters and others is essential. The prevalence of coronary artery disease will be assessed by site.
Correlation of previous cardiac examination results of patients included in the pilot study with result of Computed Tomography Angiography and Invasive Coronary Angiography | up to a maximum of 2 years after completion of pilot study at all sites
  Previous cardiac examination results will be assessed in the pilot study, reflecting the routinely performed tests before referral to Computed Tomography Angiography and Invasive Coronary Angiography. The correlation of these previous tests with the CTA or ICA results will be analysed.
Comparison of hospitalisation after Invasive Coronary Angiography in different European clinical sites | up to a maximum of 2 years after completion of pilot study at all sites
  Due to differences in clinical practice and recommendations throughout Europe, patients may be hospitalized after Invasive Coronary Angiography. Analysis will be conducted to assess this cost factor.
Assessment of non-diagnostic segments in Computed Tomography Angiography and Invasive Coronary Angiography in the pilot study | up to a maximum of 2 years after completion of pilot study at all sites
  Non-diagnostic segments can occur in Computed Tomography Angiography and Invasive Coronary Angiography. This might lead to subsequent examinations, thus indicating an important cost factor.
Assessment of major cardiovascular adverse events in the pilot study | up to a maximum of 2 years after completion of pilot study at all sites
  Occurrence of major cardiovascular adverse events within 48 hours after examination will be analyzed. As major cardiovascular adverse events may lead to subsequent examinations they represent a major cost factor.
Health related Quality of Life and Lifestyle | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Group (CTA vs ICA) differences in health-related QoL instruments (SF-12 self-rated health item, SF-12 physical component summary score, EuroQol 5d-3L and Hospital Anxiety and Depression Scale). Hypothesis: There will be no group differences in QoL at 1 year and final follow-up. We will analyse sociodemographic, lifestyle and clinical predictors of changes in QoL (SF-12 physical component and VAS) between baseline and 1 year / final follow-up, separately for men and women. Important clinical predictors include significant CAD findings during the course of the study, changes in chest pain severity (Angina class), occurrence of MICE / MACE as well as baseline risk factor status (BMI, diabetes, smoking, physical inactivity, excessive alcohol intake).
Acceptance of time trade-off question in the pilot study | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Acceptance of time trade-off question in the pilot study
Comparison of the health instruments | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Comparison of the QoL questionnaires used in the pilot and in the main study (SF-12, EuroQoL 5d-3L, Hospital Anxiety and Depression Scale, and the MacNew).
Gender differences regarding all aspects of medical history | : at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Gender differences regarding all aspects of medical history will be collected at randomization and follow-up. Data will be analysed in regards to occurrence of MACE and MICE in all genders.
Gender differences in radiation exposure and gender | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Differences in radiation exposure and gender.
Gender differences regarding Quality of Life, lifestyle and socioeconomic status | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Differences regarding QoL, lifestyle and socioeconomic status at baseline as well as in regards to changes of these factors seen at the two follow-up time points in the two randomised groups and in male and female patients with and without CAD on testing.
Gender differences in examination results | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Comparison of the examination results (rate of coronary artery disease, PCI rate adjusted for CAD prevalence, occurrence of adverse events, stress tests used, patient acceptance) in all genders.
Gender differences of coronary plaque characteristics determined by Computed Tomography | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Gender differences of coronary plaque characteristics determined by CT including parameters like coronary plaque assessment, including calcified, mixed and non-calcified plaques, remodeling index, ring-sign, spotty calcification.
Gender differences of myocardial resting blood flow / tissue characteristics determined by Computed Tomography Angiography | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Gender differences of myocardial resting blood flow / tissue characteristics determined by cardiac CT using parameters such as regional and global TPR, AD, PI, perfusion defects, myocardial calcification, myocardial fatty infiltration, myocardial thinning.
Diagnostic value of Computed Tomography in men vs women - frequency of true positive findings in patients referred for Invasive Coronary Angiography | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Diagnostic value of CT in men vs women - frequency of true positive findings in patients referred for ICA - i.e. frequency of revascularization in patients referred for ICA based on CT with and without ischemia testing, CT findings, Ischemia testing findings, ICA findings and revascularization in patients of the CT group referred to ICA as a consequence of index evaluation, radiation dose.
Gender differences of pulmonary findings of Computed Tomography Angiography | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Composite outcome: Gender differences of pulmonary findings of cardiac CT a) signs of pulmonary congestion: Ground-Glass Opacification (GGO), Pleural effusions, interlobular transudate high density pulmonary attenuation index b) pulmonary emphysema (with/without CAD), low density pulmonary attenuation index c) Pulmonary embolism (major, minor).
Gender differences of structural Computed Tomography Angiography findings | at baseline, at 1-year follow-up and final follow-up to a max of 4 years
  Gender differences of structural cardiac CT findings including parameters such as LV-mass, volumes and dimensions of Left Ventricle (LV), Left Atrium (LA), Right Ventricle (RV), Right Atrium (RA) and blood pressure.
Analysis of occurrence in Major Adverse Cardiac Events in subgroups | at baseline, at 1-year follow-up and final follow up to a max of 4 years
  Composite outcome: Analysis of occurrence in MACE as a secondary outcome in following subgroups:
  Angina classification groups CT plaque characteristic groups: high risk versus other plaques versus no plaques Gender: male versus female Age: occurrence of MACE in patient a) under 45 years, b) between 45 and 65 years and c) over 65 years QoL: patients with significant QoL reductions versus patients with no changes in QoL BMI: Patients with BMI a) under 25, b) between 25 and 30 and c) over 30
Major Adverse Cardiac Events in different composites | at baseline, at 1-year follow-up and final follow up to a max of 4 years
  Composite outcome: definition of MACE as a) vascular death or Myocardial Infarction (MI), b) cardiac death or MI.
Occurrence of Myocardial Infarction and stroke | at baseline, at 1-year follow-up and final follow up to a max of 4 years
  Occurrence of myocardial infarction and stroke

CONTACTS AND LOCATIONS:
Overall Officials: Marc Dewey, Prof. Dr., Principal Investigator — Charite University, Berlin, Germany
Locations (20):
- Medizinische Universitaet Innsbruck, Innsbruck, Austria
- Fakultni Nemocnice V Motole, Prague, Czechia
- Region Hovedstaden, Copenhagen, Denmark
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Alb Fils Kliniken Gmbh, Göppingen
  - Universitaet Leipzig, Leipzig
- Semmelweis Egyetem, Budapest, Hungary
- University College Dublin, National University of Ireland, Dublin, Ireland
- Italy (2):
  - Universita Degli Studi Di Cagliari, Cagliari
  - Universita Degli Studi Di Roma La Sapienza, Rome
- Paula Stradina Kliniska Universitates Slimnica As, Riga, Latvia
- Lietuvos Sveikatos Mokslu Universitetas, Kaunas, Lithuania
- Wojewodzki Szpital Specjalistyczny We Wroclawiu, Wroclaw, Poland
- Centro Hospitalar de Vila Nova de Gaia/Espinho Epe, Vila Nova de Gaia, Portugal
- Cardio Med Srl, Târgu Mureş, Romania
- Institut Za Kardiovaskularne Bolesti Vojvodine, Novi Sad, Serbia
- Institut Catala de La Salut, Barcelona, Spain
- United Kingdom (3):
  - South Eastern Health and Social Care Trust Nhs, Belfast
  - University of Glasgow, Glasgow
  - Aintree University Hospital Nhs Foundation Trust, Liverpool

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Napp AE, Haase R, Laule M, Schuetz GM, Rief M, Dreger H, Feuchtner G, Friedrich G, Spacek M, Suchanek V, Fuglsang Kofoed K, Engstroem T, Schroeder S, Drosch T, Gutberlet M, Woinke M, Maurovich-Horvat P, Merkely B, Donnelly P, Ball P, Dodd JD, Quinn M, Saba L, Porcu M, Francone M, Mancone M, Erglis A, Zvaigzne L, Jankauskas A, Sakalyte G, Haran T, Ilnicka-Suckiel M, Bettencourt N, Gama-Ribeiro V, Condrea S, Benedek I, Cemerlic Adjic N, Adjic O, Rodriguez-Palomares J, Garcia Del Blanco B, Roditi G, Berry C, Davis G, Thwaite E, Knuuti J, Pietila M, Kepka C, Kruk M, Vidakovic R, Neskovic AN, Diez I, Lecumberri I, Geleijns J, Kubiak C, Strenge-Hesse A, Do TH, Fromel F, Gutierrez-Ibarluzea I, Benguria-Arrate G, Keiding H, Katzer C, Muller-Nordhorn J, Rieckmann N, Walther M, Schlattmann P, Dewey M; DISCHARGE Trial Group. Computed tomography versus invasive coronary angiography: design and methods of the pragmatic randomised multicentre DISCHARGE trial. Eur Radiol. 2017 Jul;27(7):2957-2968. doi: 10.1007/s00330-016-4620-z. Epub 2016 Nov 18. PMID 27864607
- [Background] Dewey M, Rief M, Martus P, Kendziora B, Feger S, Dreger H, Priem S, Knebel F, Bohm M, Schlattmann P, Hamm B, Schonenberger E, Laule M, Zimmermann E. Evaluation of computed tomography in patients with atypical angina or chest pain clinically referred for invasive coronary angiography: randomised controlled trial. BMJ. 2016 Oct 24;355:i5441. doi: 10.1136/bmj.i5441. PMID 27777234
- [Background] Haase R, Dodd JD, Kauczor HU, Kazerooni EA, Dewey M. Developing a lung nodule management protocol specifically for cardiac CT: Methodology in the DISCHARGE trial. Eur J Radiol Open. 2020 Jun 25;7:100235. doi: 10.1016/j.ejro.2020.100235. eCollection 2020. PMID 32637465
- [Result] De Rubeis G, Napp AE, Schlattmann P, Geleijns J, Laule M, Dreger H, Kofoed K, Sorgaard M, Engstrom T, Tilsted HH, Boi A, Porcu M, Cossa S, Rodriguez-Palomares JF, Xavier Valente F, Roque A, Feuchtner G, Plank F, Stechovsky C, Adla T, Schroeder S, Zelesny T, Gutberlet M, Woinke M, Karolyi M, Karady J, Donnelly P, Ball P, Dodd J, Hensey M, Mancone M, Ceccacci A, Berzina M, Zvaigzne L, Sakalyte G, Basevicius A, Ilnicka-Suckiel M, Kusmierz D, Faria R, Gama-Ribeiro V, Benedek I, Benedek T, Adjic F, Cankovic M, Berry C, Delles C, Thwaite E, Davis G, Knuuti J, Pietila M, Kepka C, Kruk M, Vidakovic R, Neskovic AN, Lecumberri I, Diez Gonzales I, Ruzsics B, Fisher M, Dewey M, Francone M; DISCHARGE Trial Group. Pilot study of the multicentre DISCHARGE Trial: image quality and protocol adherence results of computed tomography and invasive coronary angiography. Eur Radiol. 2020 Apr;30(4):1997-2009. doi: 10.1007/s00330-019-06522-z. Epub 2019 Dec 16. PMID 31844958
- [Result] Rieckmann N, Neumann K, Feger S, Ibes P, Napp A, Preuss D, Dreger H, Feuchtner G, Plank F, Suchanek V, Veselka J, Engstrom T, Kofoed KF, Schroder S, Zelesny T, Gutberlet M, Woinke M, Maurovich-Horvat P, Merkely B, Donnelly P, Ball P, Dodd JD, Hensey M, Loi B, Saba L, Francone M, Mancone M, Berzina M, Erglis A, Vaitiekiene A, Zajanckauskiene L, Haran T, Suckiel MI, Faria R, Gama-Ribeiro V, Benedek I, Rodean I, Adjic F, Cemerlic Adjic N, Rodriguez-Palomares J, Garcia Del Blanco B, Brooksbank K, Collison D, Davis G, Thwaite E, Knuuti J, Saraste A, Kepka C, Kruk M, Benedek T, Ratiu M, Neskovic AN, Vidakovic R, Diez I, Lecumberri I, Fisher M, Ruzsics B, Hollingworth W, Gutierrez-Ibarluzea I, Dewey M, Muller-Nordhorn J. Health-related qualify of life, angina type and coronary artery disease in patients with stable chest pain. Health Qual Life Outcomes. 2020 May 14;18(1):140. doi: 10.1186/s12955-020-01312-4. PMID 32410687
- [Result] Feger S, Ibes P, Napp AE, Lembcke A, Laule M, Dreger H, Bokelmann B, Davis GK, Roditi G, Diez I, Schroder S, Plank F, Maurovich-Horvat P, Vidakovic R, Veselka J, Ilnicka-Suckiel M, Erglis A, Benedek T, Rodriguez-Palomares J, Saba L, Kofoed KF, Gutberlet M, Adic F, Pietila M, Faria R, Vaitiekiene A, Dodd JD, Donnelly P, Francone M, Kepka C, Ruzsics B, Muller-Nordhorn J, Schlattmann P, Dewey M. Clinical pre-test probability for obstructive coronary artery disease: insights from the European DISCHARGE pilot study. Eur Radiol. 2021 Mar;31(3):1471-1481. doi: 10.1007/s00330-020-07175-z. Epub 2020 Sep 9. PMID 32902743
- [Derived] Dodd JD, Bosserdt M, Oleksiak A, Vattay B, Bech Moller M, Benedek TM, Campbell F, Rodriguez-Palomares JF, Flynn S, Serna-Higuita LM, Sox H, Dewey M. Comparative Analysis of Cardiac CT and Invasive Coronary Angiography for Suspected Stable Coronary Artery Disease and Subsequent Functional Testing and Revascularization: A Prespecified Secondary DISCHARGE Randomized Trial Analysis. Radiol Cardiothorac Imaging. 2025 Aug;7(4):e240526. doi: 10.1148/ryct.240526. PMID 40874840
- [Derived] DISCHARGE Trial Group; Rieckmann N, Neumann K, Maurovich-Horvat P, Kofoed KF, Benedek T, Bosserdt M, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Adic NC, Gutberlet M, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Kubiak C, Hansen KS, Muller-Nordhorn J, Merkely B, Knudsen AD, Benedek I, Orr C, Valente FX, Zvaigzne L, Suchanek V, Zajanckauskiene L, Adic F, Woinke M, Waters D, Lecumberri I, Thwaite E, Laule M, Kruk M, Neskovic AN, Birtolo LI, Kusmierz D, Feuchtner G, Pietila M, Ribeiro VG, Drosch T, Delles C, Matta G, Fisher M, Szilveszter B, Larsen L, Ratiu M, Kelly S, Garcia Del Blanco B, Drobni ZD, Jurlander B, Regan S, Calabria HC, Boussoussou M, Engstrom T, Hodas R, Napp AE, Haase R, Feger S, Mohamed MMA, Dreger H, Rief M, Wieske V, Estrella M, Michallek F, Mark DB, Martus P, Dodd JD, Sox HC, Serna-Higuita LM, Dewey M. Health Status Outcomes After Computed Tomography or Invasive Coronary Angiography for Stable Chest Pain: A Prespecified Secondary Analysis of the DISCHARGE Randomized Clinical Trial. JAMA Cardiol. 2025 Jul 1;10(7):728-739. doi: 10.1001/jamacardio.2025.0992. PMID 40366703
- [Derived] DISCHARGE Trial Group; Bosserdt M, Serna-Higuita LM, Feuchtner G, Merkely B, Kofoed KF, Benedek T, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Adic NC, Gutberlet M, Dodd JD, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Rieckmann N, Kubiak C, Hansen KS, Muller-Nordhorn J, Szilveszter B, Sigvardsen PE, Benedek I, Orr C, Valente FX, Zvaigzne L, Suchanek V, Jankauskas A, Adic F, Woinke M, Hensey M, Lecumberri I, Thwaite E, Laule M, Kruk M, Neskovic AN, Mancone M, Kusmierz D, Pietila M, Ribeiro VG, Drosch T, Delles C, Porcu M, Fisher M, Boussoussou M, Kragelund C, Aurelian R, Kelly S, Garcia Del Blanco B, Rubio A, Maurovich-Horvat P, Hove JD, Rodean I, Regan S, Cuellar-Calabria H, Molnar L, Larsen L, Hodas R, Napp AE, Haase R, Feger S, Mohamed M, Neumann K, Dreger H, Rief M, Wieske V, Estrella M, Martus P, Sox HC, Dewey M. Age and Computed Tomography and Invasive Coronary Angiography in Stable Chest Pain: A Prespecified Secondary Analysis of the DISCHARGE Randomized Clinical Trial. JAMA Cardiol. 2024 Apr 1;9(4):346-356. doi: 10.1001/jamacardio.2024.0001. PMID 38416472
- [Derived] Mancone M, Mezquita AJV, Birtolo LI, Maurovich-Horvat P, Kofoed KF, Benedek T, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Adic NC, Gutberlet M, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Rieckmann N, Kubiak C, Hansen KS, Muller-Nordhorn J, Merkely B, Sigvardsen PE, Benedek I, Orr C, Valente FX, Zvaigzne L, Suchanek V, Jankauskas A, Adic F, Woinke M, Keane S, Lecumberri I, Thwaite E, Kruk M, Jovanovic V, Kusmierz D, Feuchtner G, Pietila M, Ribeiro VG, Drosch T, Delles C, Palmisano V, Fisher M, Drobni ZD, Kragelund C, Aurelian R, Kelly S, Del Blanco BG, Rubio A, Boussoussou M, Hove JD, Rodean I, Regan S, Calabria HC, Becker D, Larsen L, Hodas R, Napp AE, Haase R, Feger S, Mohamed M, Neumann K, Dreger H, Rief M, Wieske V, Douglas PS, Estrella M, Bosserdt M, Martus P, Serna-Higuita LM, Dodd JD, Dewey M. Impact of smoking in patients with suspected coronary artery disease in the randomised DISCHARGE trial. Eur Radiol. 2024 Jun;34(6):4127-4141. doi: 10.1007/s00330-023-10355-2. Epub 2023 Nov 22. PMID 37991508
- [Derived] DISCHARGE Trial Group; Kofoed KF, Bosserdt M, Maurovich-Horvat P, Rieckmann N, Benedek T, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Adic F, Gutberlet M, Dodd JD, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Kubiak C, Hansen KS, Muller-Nordhorn J, Merkely B, Jorgensen TS, Benedek I, Orr C, Valente FX, Zvaigzne L, Suchanek V, Zajanckauskiene L, Cankovic M, Woinke M, Keane S, Lecumberri I, Thwaite E, Laule M, Kruk M, Neskovic AN, Mancone M, Kusmierz D, Feuchtner G, Pietila M, Ribeiro VG, Drosch T, Delles C, Loi B, Fisher M, Szilveszter B, Sigvardsen PE, Ratiu M, Kelly S, Garcia Del Blanco B, Rubio A, Drobni ZD, Kragelund C, Rodean I, Regan S, Calabria HC, Boussoussou M, Engstrom T, Hodas R, Napp AE, Haase R, Feger S, Mohamed MMA, Serna-Higuita LM, Neumann K, Dreger H, Rief M, Wieske V, Estrella M, Martus P, Dewey M. Comparative effectiveness of initial computed tomography and invasive coronary angiography in women and men with stable chest pain and suspected coronary artery disease: multicentre randomised trial. BMJ. 2022 Oct 19;379:e071133. doi: 10.1136/bmj-2022-071133. PMID 36261169
- [Derived] DISCHARGE Trial Group; Maurovich-Horvat P, Bosserdt M, Kofoed KF, Rieckmann N, Benedek T, Donnelly P, Rodriguez-Palomares J, Erglis A, Stechovsky C, Sakalyte G, Cemerlic Adic N, Gutberlet M, Dodd JD, Diez I, Davis G, Zimmermann E, Kepka C, Vidakovic R, Francone M, Ilnicka-Suckiel M, Plank F, Knuuti J, Faria R, Schroder S, Berry C, Saba L, Ruzsics B, Kubiak C, Gutierrez-Ibarluzea I, Schultz Hansen K, Muller-Nordhorn J, Merkely B, Knudsen AD, Benedek I, Orr C, Xavier Valente F, Zvaigzne L, Suchanek V, Zajanckauskiene L, Adic F, Woinke M, Hensey M, Lecumberri I, Thwaite E, Laule M, Kruk M, Neskovic AN, Mancone M, Kusmierz D, Feuchtner G, Pietila M, Gama Ribeiro V, Drosch T, Delles C, Matta G, Fisher M, Szilveszter B, Larsen L, Ratiu M, Kelly S, Garcia Del Blanco B, Rubio A, Drobni ZD, Jurlander B, Rodean I, Regan S, Cuellar Calabria H, Boussoussou M, Engstrom T, Hodas R, Napp AE, Haase R, Feger S, Serna-Higuita LM, Neumann K, Dreger H, Rief M, Wieske V, Estrella M, Martus P, Dewey M. CT or Invasive Coronary Angiography in Stable Chest Pain. N Engl J Med. 2022 Apr 28;386(17):1591-1602. doi: 10.1056/NEJMoa2200963. Epub 2022 Mar 4. PMID 35240010
- See also: Project homepage — http://www.dischargetrial.eu
- See also: European Commission Project homepage — https://cordis.europa.eu/project/rcn/110447/factsheet/en